CLINICAL TRIAL: NCT03688555
Title: A Randomized, Double-blind, Placebo-controlled, 12-week Treatment Study to Evaluate the Effect of ACT-774312 in Subjects With Bilateral Nasal Polyposis
Brief Title: A Study to Evaluate the Effect of ACT-774312 in Subjects With Bilateral Nasal Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID-084A201; 2018-000851-42 (EudraCT Number)
Record Dates: First submitted 2018-09-18; First posted 2018-09-28 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Bilateral Nasal Polyposis
MeSH Terms: interventions — ACT-774312

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-774312 (Experimental): Participants will receive ACT-774312 (400 mg twice daily) in the morning and evening with or without food for 12 weeks together with mometasone furoate nasal spray.
  Interventions: Drug: ACT-774312
- Placebo (Placebo Comparator): Participants will receive placebo twice daily in the morning and evening with or without food for 12 weeks together with mometasone furoate nasal spray.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-774312 — ACT-774312 will be available as hard gelatin capsules containing 200 mg of ACT-774312
  Arms: ACT-774312
Drug: Placebo — Matching placebo hard gelatin capsules
  Arms: Placebo

SUMMARY:
The study will evaluate the effect of ACT-774312 on the nasal polyps and will assess the safety and tolerability of ACT-774312 in the patients with bilateral nasal polyposis

DETAILED DESCRIPTION:
The clinical trial has 3 periods:

Screening and run-in period (4 Weeks). This period starts with the screening visit, and ends on Day 1, just before the first study treatment administration. At Visit 1, all participants will enter a run-in period of 4 weeks on mometasone furoate nasal spray of 2 actuations (50 μg per actuation) in each nostril twice daily (total daily dose of 400 μg), unless they were intolerant to twice daily intranasal corticosteroids, in which case they could use a lower dose regimen, i.e., 200 μg once daily.

Treatment period (ACT-774312 or placebo for 12 weeks). This period will start on Day 1 with the first administration of study treatment and consists of 4 visits: Week 2, Week 4, Week 8, and Week 12. Provided that the nasal polyp score (NPS) does not change during the run-in period, participants will be randomized to ACT-774312 (400 mg twice daily) or placebo (twice daily) for 12 weeks. During the double-blind randomized treatment all participants will continue with mometasone furoate nasal spray background therapy.

Post-treatment period (4 Weeks). This period will start after the Week 12 Visit and end at Week 16 (End-of-Study).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study mandated procedure.
* A minimum bilateral nasal polyp score (NPS) of 5 out of a maximum of 8 for both nostrils (with at least a score of 2 for each nostril) despite completion of a prior intranasal corticosteroids (INCS) treatment for at least 8 weeks before screening, with at least the 6 last weeks on INCS spray.
* Presence of at least 2 of the following symptoms at screening:

  * nasal blockade/obstruction
  * nasal discharge (anterior/posterior nasal drip)
  * reduction or loss of smell.
* Male and female participants aged between 18 and 70 years (inclusive) at screening.
* Systolic blood pressure 90 to 160 mmHg, diastolic blood pressure 50 to 100 mmHg, pulse rate 45 to 100 bpm (inclusive), measured on the dominant arm, after 5 minutes in the supine position at screening.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test pre-dose on Day 1. Women of childbearing potential must consistently and correctly use (from at least first dosing, during the entire study, and for at least 30 days after last study treatment intake) 1 highly effective method of contraception with a failure rate of less than 1% per year, be sexually abstinent, or have a vasectomized partner. Hormonal contraceptive must have been initiated at least 1 month before first study treatment administration.

Exclusion Criteria:

* CYP2C9 poor metabolizer.
* Participant with severe renal function impairment (≤ 29 mL/min/1.73 m2) which is defined by estimated glomerular filtration rate at screening using the Modification of Diet in Renal Disease (MDRD) formula.
* Participant with Sino-Nasal Outcome Test (SNOT-22) less than 20.
* Participant who has required oral corticosteroids (OCS) within the 2 months before screening or is scheduled to receive OCS during the study period for another condition.
* Participant who has required INCS drops within the 6 weeks before screening.
* Participant who was injected with long-lasting activity corticosteroids within the 3 months before screening or is scheduled to receive these during the study period for another condition.
* Participant who has undergone any nasal surgery within 6 months before screening.
* Participant with conditions/concomitant diseases making them non-evaluable for the primary efficacy endpoint such as:

  * Antrochoanal polyps
  * Nasal septal deviation that occludes at least one nostril
  * Acute sinusitis, nasal infection or upper respiratory infection at screening or in the 2 weeks before screening
  * Ongoing rhinitis medicamentosa
  * Churg-Strauss syndrome, Young's syndrome, Kartagener's syndrome or dyskinetic ciliary syndromes, Cystic fibrosis
  * Signs or a CT scan suggestive of Allergic fungal rhinosinusitis.
* Participants with co-morbid asthma are excluded if:

  * Forced expiratory volume in one second (FEV1) ≤ 60% of predicted normal OR
  * An exacerbation requiring systemic (oral and/or parenteral) steroid treatment or hospitalization (>24 h) for treatment of asthma has occurred within 3 months prior screening OR
  * They are on a dose higher than 1000 μg fluticasone or the equivalent of inhaled corticosteroids (ICS).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Participants with active autoimmune disease (e.g., Hashimoto's thyroiditis, Graves' disease, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, psoriasis vulgaris, rheumatoid arthritis).
* Participant considered as vulnerable (e.g., sponsor or site employee, investigator subordinate, participant incapable of giving consent, participant committed to an institution by way of official or judicial order).
* Participant with liver injury related criteria:

  * Underlying hepatobiliary disease OR
  * Alanine aminotransferase greater than 3 x upper limit of normal, OR
  * or Bilirubin greater than 2 x upper limit of normal.
* Participant with unstable NPS during the run-in period, i.e. altered score at Day 1 when compared to the screening NPS (assessed locally by the investigator).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (2):
- University Hospital Ghent, Ghent, Belgium
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between the 19 Oct 2018 and 01 Dec 2020. The study was conducted at 2 sites in 2 countries (Belgium and Germany), both sites randomized participants.
Pre-assignment Details: At screening, patients were on a stable regimen of intranasal corticosteroids (INCS) for at least 8 weeks. If a participant was using an INCS product different from mometasone furoate nasal spray prior to the screening visit, the investigator had to switch to mometasone furoate nasal spray at screening (Visit 1). Only once a participant was eligible for randomization was data collected.
Groups:
- Mometasone Furoate: All participants were placed on non-investigational, standard background therapy: Mometasone furoate nasal spray 50 μg/actuation nasal spray, suspension for 4 weeks (Visit 1 to Visit 2). Dosing regimen: 2 actuations (50 μg/actuation) in each nostril twice daily (or once daily if twice daily was not tolerated).
- ACT-774312: Participants received ACT-774312 400 mg twice daily in the morning and evening with or without food for 12 weeks. In addition, participants also continued with their standard background therapy of mometasone furoate nasal spray.
- Placebo: Participants received matching placebo hard gelatin capsules twice daily in the morning and evening with or without food for 12 weeks. In addition, participants also continued with their standard background therapy of mometasone furoate nasal spray.
Period: Run-in Period
Arm/Group | Mometasone Furoate | ACT-774312 | Placebo
Started | 10 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Mometasone Furoate | ACT-774312 | Placebo
Started | 0 (All 10 participants that completed the run-in period were eligible to be randomized to ACT-774312 or placebo.) | 7 | 3
Completed | 0 | 7 | 2
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis set included all randomized participants who received at least one dose of the study treatment. Participants were evaluated according to the actual study treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT-774312 | Placebo | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.9) | 54.7 (5.5) | 51.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 2 | 1 | 3
  Germany | 5 | 2 | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram(s)/square meter] | 28.2 (5.25) | 26.0 (2.81) | 27.5 (4.61)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Nasal Polyp Score as Measured by Nasal Endoscopy (Assessed Centrally)
Description: Independent reviewers, blinded to treatment, reviewed image recordings of nasal endoscopies to determine total endoscopic nasal polyp score based on nasal polyp size. The right and left nostrils were scored from 0 to 4 (0 = No polyps; 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle concha; 2 = Polyps reaching below the lower border of the middle turbinate; 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle concha; and 4 = Large polyps causing complete obstruction/congestion of the inferior meatus). The total score is the sum of the right and left nostril scores and ranges from 0 to 8, higher scores indicate greater disease severity. Data up to Week 12 were included in the analyses. The Day 1 value was the baseline. Change from Baseline = (Post-baseline visit value) minus (Baseline visit value). A negative change indicates worsening.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: Per-protocol set. This analysis set includes all randomized participants who completed the treatment up to Week 12 without protocol deviations that may affect the evaluation of the primary endpoints.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- ACT-774312: Participants received ACT-774312 (400 mg twice daily) in the morning and evening with or without food for 12 weeks. In addition, participants also continued with their standard background therapy of mometasone furoate nasal spray.
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale | -0.23 (0.161) | -0.99 (0.253)
Statistical Analysis 1: Comparison: ACT-774312 vs Placebo; Test type: Superiority; p = 0.062, Mixed model for repeated measurements — All Nasal Polyp Score (NPS) values observed between baseline and Week 12 were included in the analysis. Changes from baseline to post-baseline visits in NPS were analyzed using a Mixed Model for Repeated Measurement (MMRM); LS means difference = 0.76, 95% CI 2-sided [-0.06 to 1.59], Standard Error of Mean 0.301

2. Secondary Outcome: Change From Baseline to Week 12 in Sinus Opacifications as Assessed by Computed Tomography Scan Using the Modified Lund Mackay Score (Assessed Centrally)
Description: Independent blinded reviewers reviewed image recordings of the computed tomography scan. The modified Lund Mackay Score scores were given for the degree of opacification and their location in the sinus. The right and left sinuses are divided into 6 portions, i.e., maxillary sinus, anterior ethmoid sinuses, posterior ethmoid sinuses, sphenoid sinus, frontal sinus, and ostiomeatal complex (OMC). The OMC is given a score of 0 (no obstruction) or 1 (obstruction) for the frontal recess, middle meatus, infundibulum, and the sphenoethmoidal recess channels. The total score is the sum of the right and left nostril scores and range from 0 to a maximum of 48. A positive change from baseline (Day 1) indicates a worsening.
  Change in the modified Lund-Mackay score = modified Lund-Mackay score at Week 12 minus the modified Lund-Mackay score at baseline.
  A positive change from baseline indicated a worsening in the modified Lund-Mackay Score at Week 12 compared to baseline.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale | 0.86 (1.24) | 4.84 (1.96)
Statistical Analysis 1: Comparison: ACT-774312 vs Placebo; Test type: Superiority; p = 0.161, ANCOVA; LS means difference = -3.98, 95% CI 2-sided [-10.41 to 2.45], Standard Error of Mean 2.316

3. Secondary Outcome: Change From Baseline to Week 12 in the Volume of Air in the Left Maxillary Sinus
Description: Independent reviewers, blinded to treatment, reviewed image recordings of the computed tomography scan and performed 3D volumetric measurements of the left maxillary sinus. Absolute changes from baseline were calculated for volume of air (mL). Change in 3D volumetric measurement = (3D volumetric measurement at Week 12) minus (3D volumetric measurement at baseline). A positive change from baseline indicates that more volume for air is in the left maxillary sinus since the baseline visit. More volume of air indicates that the polyposis is improving in the left maxillary sinus.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter(s)
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
milliliter(s) | 1.17 (1.72) | -1.08 (2.48)

4. Secondary Outcome: Change From Baseline to Week 12 in the Volume of Air in the Right Maxillary Sinus
Description: Independent reviewers, blinded to treatment, reviewed image recordings of the computed tomography scan and performed 3D volumetric measurements of the right maxillary sinus. Absolute changes from baseline were calculated for the volume of air (mL) in the right maxillary sinus: Change in 3D volumetric measurement = (3D volumetric measurement at Week 12) minus (3D volumetric measurement at baseline). A positive change from baseline indicates that more volume for air is in the right maxillary sinus since the baseline visit. More volume of air indicates that the polyposis is improving in the right maxillary sinus.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter(s)
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
milliliter(s) | -0.94 (4.36) | 1.77 (1.34)

5. Secondary Outcome: Change From Baseline to Week 12 in the Left Maxillary Sinus Mucosal Volume
Description: Independent reviewers, blinded to treatment, reviewed image recordings of the computed tomography scan and performed 3D volumetric measurements of the left maxillary sinus. Absolute changes from baseline were calculated for the volume of air (mL) in the left maxillary sinus: Change in 3D volumetric measurement = (3D volumetric measurement at Week 12) minus (3D volumetric measurement at baseline). A negative change from baseline indicates that the left maxillary sinus mucosal volume has decreased since the baseline visit. More mucosal volume, a positive change, indicates that the polyposis is worsening in the left maxillary sinus.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter(s)
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
milliliter(s) | -1.72 (1.72) | -1.08 (2.48)

6. Secondary Outcome: Change From Baseline to Week 12 in the Right Maxillary Sinus Mucosal Volume
Description: Independent reviewers, blinded to treatment, reviewed image recordings of the computed tomography scan and performed 3D volumetric measurements of the right maxillary sinus. Absolute changes from baseline were calculated for the volume of air (mL) in the right maxillary sinus: Change in 3D volumetric measurement = (3D volumetric measurement at Week 12) minus (3D volumetric measurement at baseline). A negative change from baseline indicates that the right maxillary sinus mucosal volume has decreased since the baseline visit. More mucosal volume, a positive change, indicates that the polyposis is worsening in the right maxillary sinus.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter(s)
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
milliliter(s) | 0.94 (4.36) | -1.78 (1.34)

7. Secondary Outcome: Change From Baseline to Week 12 in the University of Pennsylvania Smell Identification Test
Description: The UPSIT (University of Pennsylvania Smell Identification Test) is a test that measures an individual's ability to detect odors. It consists of 4 workbooks of 10 pages each. On each page there is a different "scratch and sniff" strip which is embedded with a micro-encapsulated odorant and a question regarding the smell detected with a four-choice option for the response. The total number of questions in the UPSIT is 40. The number of correct responses regarding the smells being experienced is summed to provide a total score that ranges from 0 to 40, with a higher score indicating a better sense of smell.
  Absolute changes from baseline to Week 12 was calculated as follows: Change in UPSIT score = (UPSIT score at Week 12) minus (UPSIT score at baseline). A positive change from baseline in the UPSIT score is considered a favorable outcome.
Time Frame: Pre-dose (Baseline on Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale | 1.0 (8.4) | -0.5 (0.7)

8. Secondary Outcome: Change From Baseline in the Visual Analog Scale Symptoms Score
Description: The participant was asked to score on a Visual Analog Scale (VAS) the answer to the question: "How troublesome are your symptoms?" (for the 5 following symptoms: nasal obstruction, nasal discharge, mucus in the throat, loss of smell, facial pain). The VAS ranges from 0 (Not at all troublesome) to 100 (Extremely troublesome). The sum of the score of all symptoms were added to a total VAS score which ranged from 0 to 500. The higher the VAS score the more troublesome the symptoms. Absolute changes from baseline to Weeks 2, 4, 8, 12, and End of Study are calculated as follows: Change in total VAS score = Change in total VAS score = (Total VAS score at visit) minus (Total VAS score at baseline). A negative change from baseline indicates an improvement.. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12 and Week 16 (End-of-Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale
  Baseline | 304.0 (75.0) | 323.5 (95.5)
  Change from baseline at Week 2 | -69.8 (68.4) | -77.5 (136.5)
  Change from baseline at Week 4 | -108.0 (106.0) | -58.0 (18.4)
  Change from baseline at Week 8 | -70.5 (121.3) | -88.5 (61.5)
  Change from baseline at Week 12 | -90.0 (55.9) | -156.0 (123.7)
  Change from baseline at Week 16 (End-of-Study) | -105.4 (78.9) | -57.0 (104.7)

9. Secondary Outcome: Physician Global Assessment of Change in Disease Severity
Description: The Physician Global Assessment of Disease Severity questionnaire (PGAC-DS) was completed by the physician at Visit 2 and at each subsequent site visit until the End-of-Study (Week 16). The PGAC-DS questionnaire is a self-administered 1-item questionnaire designed to assess the physician's impression of change in disease severity since study treatment start. The physician rated the change since the participant study treatment start. The physician rated the change since the participant started study treatment on a 7-point scale. The rating for the overall score is: 'very much improved' (is scored 1), 'much improved' (is scored 2), 'minimally improved' (is scored 3), 'no change' (is scored 4), 'minimally worse' (is scored 5), 'much worse' (is scored 6), or 'very much worse' (is scored 7).
Time Frame: Week 2, Week 4, Week 8, Week 12, and Week 16 (End-of-Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale
  Week 2 | 3.4 (0.5) | 3.0 (1.4)
  Week 4 | 3.0 (0.7) | 3.0 (1.4)
  Week 8 | 3.6 (1.3) | 2.5 (0.7)
  Week 12 | 3.4 (0.5) | 4.0 (1.4)
  Week 16 (End-of-Study) | 3.6 (0.5) | 4.0 (1.4)

10. Secondary Outcome: Change From Baseline in the Sino-Nasal Outcome Test
Description: SNOT-22 (Sino-Nasal Outcome Test) is a disease specific quality of life questionnaire measure that comprises a list of 22 symptoms and social or emotional consequences of the nasal disorder. Every participant was asked to rate how severe each problem had been for them over the past 2 weeks on a scale from 0 (no problem) to 5 (problem as bad as it can be). The total score is the sum of the scores for all 22 items, ranging from 0 to 110. Higher total scores on the SNOT-22 imply greater impact on Quality of Life. Absolute changes from baseline to Weeks 2, 4, 8, 12, and 16 were calculated as follows: Change in SNOT-22 score = (SNOT-22 score at visit) minus (SNOT-22 score at baseline). A negative change from baseline in SNOT-22 is considered a favorable outcome.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, and Week 16 (End-of-Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants received matching placebo hard gelatin capsules twice daily in the morning and evening with or without food for 12 weeks.In addition, participants also continued with their standard background therapy of mometasone furoate nasal spray.
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale
  Baseline | 61.4 (9.2) | 59.5 (19.1)
  Change from baseline at Week 2 | -7.2 (18.5) | -22.5 (27.6)
  Change from baseline at Week 4 | -21.4 (11.0) | -21.5 (16.3)
  Change from baseline at Week 8 | -14.4 (14.7) | -29.0 (18.4)
  Change from baseline at Week 12 | -15.2 (5.3) | -21.5 (16.3)
  Change from baseline at Week 16 (End-of-Study) | -16.4 (3.9) | -24.0 (22.6)

11. Secondary Outcome: Patient Global Impression of Change in Disease Severity
Description: A patient global impression of change in disease severity questionnaire (PGIC-DS) was completed by the participant at Week 2 and at each subsequent site visit until the End-of-study visit. The PGIC-DS questionnaire was a self-administered 1-item questionnaire designed to assess participant's impression of change in disease severity since study treatment start. Participants rated their change since they started study treatment for the overall severity of the disease symptoms on a 7-point scale (1 to 7) scored as: "very much improved" (1),"much improved," (2), "minimally improved,"(3) "no change," (4) "minimally worse," (5) "much worse," (6) or "very much worse" (7).
Time Frame: Week 2, Week 4, Week 8, Week 12, and Week 16 (End-of-Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACT-774312 | Placebo
Number analyzed (Participants) | 5 | 2
score on a scale
  Week 2 | 3.2 (0.4) | 2.5 (2.1)
  Week 4 | 3.0 (0.7) | 2.5 (2.1)
  Week 8 | 3.4 (1.5) | 2.0 (0.0)
  Week 12 | 3.4 (0.5) | 2.0 (0.0)
  Week 16 (End-of-Study) | 3.4 (0.9) | 2.5 (0.7)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were all adverse events that occurred after first study treatment administration on Day 1 through to last study treatment administration on Day 84, and in the post-treatment period up to the end-of-study visit on Day 112.
Arm/Group | ACT-774312 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 5/7 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT-774312 (N=7) | Placebo (N=3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) — Episodes of worsening of nasal polyps.
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Worsening of asthma bronchiales.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Premenstrual headache (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 1 (1)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was initially planned as a single-center study. The protocol had to be updated accordingly for approvals for the second site in Germany.

The p-values need to be cautiously interpreted due to the small study population size.

Recruitment was put on hold on during the COVID-19 pandemic from 30 March to 28 May 2020 in Germany and from 31 March 2020 to 11 June 2020 in Belgium. Recruitment was subsequently restarted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Idorsia for review at least 30 days prior to submission for publication or presentation. Upon review, Idorsia may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03688555/Prot_SAP_000.pdf